CLINICAL TRIAL: NCT04862130
Title: Rehabilitative Evaluation of Functional Abilities in Children/Adolescents Affected by Cancer: a Validation Study of the GMFM-88 Scale and of the Functional Abilities Assessment in Pediatric Oncology (FAAP-O) Scale
Brief Title: Validation of the GMFM-88 Scale and of the FAAP-O Scale in Pediatric Patients Affected by Cancer
Acronym: FAAP-O
Status: Completed | Type: Observational
Sponsor: Associazione Italiana Ematologia Oncologia Pediatrica (Other)
Responsible Party: Sponsor
Other Study IDs: FAAP-O
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Oncology
Keywords: Physiotherapy; Rehabilitation; Functional abilities evaluation; motor function evaluation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to validate the Gross Motor Function Measure Scale-88 (GMFM-88) on the Italian pediatric cancer population. The secondary objective is to implement the use of the GMFM-88 in clinical practice by validating a reduced panel of items that will be called the Functional Ability Assessment in Pediatric Oncology (FAAP-O) Scale.

DETAILED DESCRIPTION:
In recent decades, improvements in the treatment of pediatric cancer patients have resulted in increased survival rates. Consequentially, clinicians now pay more attention to the quality of life of these patients, both during and after treatment. Functional abilities have an important role in the quality of life and these skills can be compromised by the tumor itself or by anti-neoplastic treatments. A recent Cochrane review regarding rehabilitation and motor activity in this population has documented the effectiveness of exercise in children with cancer. Furthermore, to improve the rehabilitation care of pediatric cancer patients it is important to broaden the research by structuring multi-center trials, which allow the collection of longitudinal data. Objective, repeatable, specific, and sensitive rehabilitation assessment tools are needed, to define the functional status of the patient and to measure the motor outcomes. The psychometric properties of a measurement are closely linked to the specific population in which the measurement is used. Currently, there are two validated assessment tools for children/adolescents with cancer used to evaluate functional abilities: The Gross Motor Function Scale-Acute Lymphoblastic Leukemia (GMFM-ALL) and the Motor Performance in Pediatric Oncology (MOON). The ladder has the merit of being structured to evaluate the motor skills of children/adolescents affected by various forms of cancer but it also presents some limits. This test does not investigate functional abilities in a rehabilitation optic and it requires the use of specific materials that can reduce its usability in multicenter trials. The GMFM-ALL scale is a modified version of the Gross Motor Function Measure 88 (GMFM-88) Scale. This scale is specific only for children/adolescents with Lymphoblastic Leukemia and it mainly evaluates motor skills that require a high functional level (i.e. jumps, running), possessed neither by younger children nor by those who show major physical impairments or during specific phases of cancer treatment, such as palliative care.

The GMFM-88 scale is a rehabilitation assessment tool that was originally created to investigate functional abilities in children affected by cerebral palsy (CP) and has subsequently been validated for other populations of pediatric patients. It was also used to evaluate functional abilities in some studies conducted on pediatric cancer patients. Some aspects make this tool easily applicable in multicenter studies: it does not require any material to be administered nor a specific certified training to use it and, lastly, it comprises all principal motor skills including the basic ones (i.e. lying and rolling on the ground).

ELIGIBILITY:
Inclusion Criteria:

* age between 6 months - 17 years and 11 months
* diagnosis of oncological disease
* being during antineoplastic treatment or up to 1 year off-therapy
* Written informed consent from patient or parents/legal representative, and age-appropriate assent.

Exclusion criteria:

• Patients that are not able and willing to comply with study visits and procedures.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents affected by cancer referred to the rehabilitation services of the participants centres.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Construct validity of the GMFM-88 in measuring functional abilities of children and adolescents affected by cancer. | up to 1 year
  Cronbach's alpha. A satisfactory index of a scale's homogeneity should have an alpha coefficient between 0.70 and 0.95.

SECONDARY OUTCOMES:
Content validity of the GMFM-88 items in evaluating functional abilities of children and adolescents affected by cancer | up to 1 year
  Content Validity Ratio (CVR). CVR values range from -1 to +1. A satisfactory CVR should be ≥ 0.70.
Construct validity of the FAAP-O in assessing functional abilities of children and adolescents affected by cancer | up to 18 months
  Cronbach's alpha A satisfactory index of a scale's homogeneity should have an alpha coefficient between 0.70 and 0.95.
Inter-observer reliability and intra-observer reliability of the FAAP-O | through study competition, an average of 2 years
  Interclass Correlation (ICC) ICC values range from 0 to 1. The repeatability of a test is considered high when ICC value is ≥ 0.8.
Test-retest reliability of the FAAP-O | through study competition, an average of 2 years
  Interclass Correlation (ICC) ICC values range from 0 to 1. The repeatability of a test is considered high when ICC value is ≥ 0.8

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Rossi, dr, Principal Investigator — A.O.U. Città della Salute e della Scienza - OIRM, Turin, Italy
Locations (10):
- Italy (10):
  - IRCCS E. Medea La Nostra Famiglia, Bosisio Parini, Lecco
  - IRCCS E. Medea La Nostra Famiglia, Conegliano, Treviso
  - Ospedale Papa Giovanni XXIII, UOS Onco-ematologia Pediatrica, Bergamo
  - Ospedale Azienda Sanitaria dell'Alto Adige - Comprensorio di Bolzano Servizio di Riabilitazione Fisica, Bolzano
  - IRCCS E. Medea La Nostra Famiglia, Brindisi
  - AOU Meyer - UP Riabilitazione, Florence
  - IRCCS Istituto Giannina Gaslini - U.O. Med Fisica e riabilitazione, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori - S.C. Cure palliative, Terapia del Dolore e Riabilitazione, Milan
  - A.O.U. Città della Salute e della Scienza - OIRM, Torino
  - IRCCS Materno Infantile Burlo Garofolo - S.C. Oncoematologia, Trieste

REFERENCES:
- [Background] De Angelis R, Sant M, Coleman MP, Francisci S, Baili P, Pierannunzio D, Trama A, Visser O, Brenner H, Ardanaz E, Bielska-Lasota M, Engholm G, Nennecke A, Siesling S, Berrino F, Capocaccia R; EUROCARE-5 Working Group. Cancer survival in Europe 1999-2007 by country and age: results of EUROCARE--5-a population-based study. Lancet Oncol. 2014 Jan;15(1):23-34. doi: 10.1016/S1470-2045(13)70546-1. Epub 2013 Dec 5. PMID 24314615
- [Background] Braam KI, van der Torre P, Takken T, Veening MA, van Dulmen-den Broeder E, Kaspers GJ. Physical exercise training interventions for children and young adults during and after treatment for childhood cancer. Cochrane Database Syst Rev. 2016 Mar 31;3(3):CD008796. doi: 10.1002/14651858.CD008796.pub3. PMID 27030386
- [Background] Byer L, Kline C, Mueller S. Clinical trials in pediatric neuro-oncology: what is missing and how we can improve. CNS Oncol. 2016 Oct;5(4):233-9. doi: 10.2217/cns-2016-0016. Epub 2016 Sep 12. PMID 27616346
- [Background] Corr AM, Liu W, Bishop M, Pappo A, Srivastava DK, Neel M, Rao B, Wilson T, Ness KK. Feasibility and functional outcomes of children and adolescents undergoing preoperative chemotherapy prior to a limb-sparing procedure or amputation. Rehabil Oncol. 2017 Jan;35(1):38-45. PMID 28948112
- [Background] Gatta G, Botta L, Rossi S, Aareleid T, Bielska-Lasota M, Clavel J, Dimitrova N, Jakab Z, Kaatsch P, Lacour B, Mallone S, Marcos-Gragera R, Minicozzi P, Sanchez-Perez MJ, Sant M, Santaquilani M, Stiller C, Tavilla A, Trama A, Visser O, Peris-Bonet R; EUROCARE Working Group. Childhood cancer survival in Europe 1999-2007: results of EUROCARE-5--a population-based study. Lancet Oncol. 2014 Jan;15(1):35-47. doi: 10.1016/S1470-2045(13)70548-5. Epub 2013 Dec 5. PMID 24314616
- [Background] Gemus M, Palisano R, Russell D, Rosenbaum P, Walter SD, Galuppi B, Lane M. Using the gross motor function measure to evaluate motor development in children with Down syndrome. Phys Occup Ther Pediatr. 2001;21(2-3):69-79. PMID 12029855
- [Background] Gohar SF, Comito M, Price J, Marchese V. Feasibility and parent satisfaction of a physical therapy intervention program for children with acute lymphoblastic leukemia in the first 6 months of medical treatment. Pediatr Blood Cancer. 2011 May;56(5):799-804. doi: 10.1002/pbc.22713. Epub 2011 Jan 16. PMID 21370414
- [Background] Gotte M, Kesting S, Albrecht C, Worth A, Bos K, Boos J. MOON-test - determination of motor performance in the pediatric oncology. Klin Padiatr. 2013 May;225(3):133-7. doi: 10.1055/s-0033-1343411. Epub 2013 Apr 18. PMID 23599231
- [Background] Lucia A, Ramirez M, San Juan AF, Fleck SJ, Garcia-Castro J, Madero L. Intrahospital supervised exercise training: a complementary tool in the therapeutic armamentarium against childhood leukemia. Leukemia. 2005 Aug;19(8):1334-7. doi: 10.1038/sj.leu.2403799. No abstract available. PMID 15931268
- [Background] Ruck-Gibis J, Plotkin H, Hanley J, Wood-Dauphinee S. Reliability of the gross motor function measure for children with osteogenesis imperfecta. Pediatr Phys Ther. 2001 Spring;13(1):10-7. PMID 17053645
- [Background] Wright MJ, Halton JM, Martin RF, Barr RD. Long-term gross motor performance following treatment for acute lymphoblastic leukemia. Med Pediatr Oncol. 1998 Aug;31(2):86-90. doi: 10.1002/(sici)1096-911x(199808)31:23.0.co;2-v. PMID 9680932
- [Derived] Rossi F, Valle M, Carlucci G, Tofani M, Galeoto G, Berchialla P, Sciannameo V, Clari M, Cardano M, Nota F, Bertin D, Calcagno A, Casalaz R, Cerboneschi M, Cervo M, Cornelli A, Fave MD, Esposito M, Ferrarese M, Imazio P, Lorenzon M, Longo L, Naretto G, Orsini N, Panzeri D, Pellegrini C, Peranzoni M, Picone F, Rabusin M, Trabacca A, Zigrino C, Martinuzzi A, Fagioli F, Ricci F. Development of Functional Abilities Assessment in Paediatric Oncology (FAAP-O) Scale for Children and Adolescents Affected by Cancer. Children (Basel). 2025 Sep 1;12(9):1163. doi: 10.3390/children12091163. PMID 41007028